CLINICAL TRIAL: NCT06369233
Title: Clinical Study to Evaluate the Anti-adhesion Efficacy and Safety of MegaShield®-SP in Comparison With Guardix-SP Plus After Spine Surgery: A Multicenter, Randomized, Subjects-independent Evaluator Blinded, Active-control Comparative, Non-inferior, Prospective Confirmatory Clinical Study
Brief Title: Clinical Study to Evaluate the Anti-adhesion Efficacy and Safety of MegaShield®-SP in Comparison With Guardix-SP Plus After Spine Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: L&C Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LNC-MS-002
Record Dates: First submitted 2024-04-12; First posted 2024-04-16 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Herniation, Disc
Keywords: disc herniation; laminectomy; anti-adhesion; disc resection; MegaShield; MegaShield-SP
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MegaShield®-SP (Experimental): The study group is applied with MegaShield®-SP after Lumbar discectomy or laminectomy. Afterwards, they visit at 2 weeks, 12 week to conduct examinations and assess Questionnaires.
  Interventions: Device: MegaShield®-SP
- Guardix-SP Plus (Active Comparator): The study group is applied with Guardix-SP after Lumbar discectomy or laminectomy. Afterwards, they visit at 2 weeks, 12 week to conduct examinations and assess Questionnaires.
  Interventions: Device: Guardix-SP Plus

INTERVENTIONS:
Device: MegaShield®-SP — MegaShield®-SP application Lumbar discectomy or laminectomy
  Arms: MegaShield®-SP
Device: Guardix-SP Plus — Guardix-SP Plus application Lumbar discectomy or laminectomy
  Arms: Guardix-SP Plus

SUMMARY:
This study is Interventional, Parallel, Double-blinded, Randomized study. Subjects aged 20 to 70 years who had a Lumbar discectomy or laminectomy, MegaShield-SP® and Guardix-SP Plus will be applied.

DETAILED DESCRIPTION:
To evaluate preventing adhesion, the study group is compared with MegaShield®-SP or Guardix-SP Plus after Lumbar discectomy or laminectomy. Afterwards, they visit at 2 weeks, 12 weeks to conduct examinations and assess Questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 to 70 years.
* Patient diagnosed with single-level lumbar disc herniation and scheduled to perform Lumbar discectomy, or patients diagnosed with single-level spinal stenosis and scheduled to perform laminectomy.
* Patients who voluntarily decide to participate in the study and voluntarily agree in writing to the informed consent form.

Exclusion Criteria:

* Patients diagnosed with multi-level lumbar disc herniation or lumbar disectomy ,far lateral lumbar disc herniation(FLLDH).
* Patient diagnosed with spinal cord disease
* Patient who needs spinal fusion
* Patient who has previous experience in spinal surgery
* Patient diagnosed with a serious liver or kidney disease
* Patients with lymph fluid or blood clotting disorder or taking antithrombotic or antiplatelet agents
* Patients with uncontrolled diabetes that may affect surgery or postoperative progress according to the investigator's judgment,
* Patients with immunocompromised or autoimmune diseases such as rheumatoid arthritis or systemic erythematosus lupus, and severe systemic immune disease
* Patients with infectious diseases or healing disorders that can interfere with the normal healing process after surgery
* Patients who received steroid epidural injections within 2 weeks from the date of screening or who took oral steroids within 24 hours
* Patients who participated in other clinical trials within 30 days from the date of screening
* Patients who are unable to take MRI scans
* Pregnant or lactating women
* Patients who are not eligible for clinical trials according to the investigator's judgement
* Patients with a history of hypersensitivity to the main and other components of the investigational device
* Patients who are scheduled to receive myelogram or lumbar puncture within 24 hours from the application of the investigational device

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
MRI scar score | At 12 weeks after surgery
  Primary effectiveness endpoint (0~4, low Scar score through MRI means better)

SECONDARY OUTCOMES:
Oswestry Disability Index(ODI) score | Before surgery, At 2, 12 weeks after surgery
  Secondary effectiveness endpoint (0~50, low ODI score means better)
Visual Analog Scale(VAS) Back & Leg Pain Score | Before surgery, At 2, 12 weeks after surgery
  Secondary effectiveness endpoint (0~100, low VAS score means better)

CONTACTS AND LOCATIONS:
Overall Officials: Siyoung Park, Principal Investigator — Yonsei University College of Medicine, Severance Hospital; Jiwon Kwon, Principal Investigator — Yonsei University College of Medicine Gangnam severance Hospital; Hojung Kim, Principal Investigator — Seoul National University Bundang Hospital; HyungYul Park, Principal Investigator — Eunpyeong St. Mary's Hospital
Locations (4):
- South Korea (4):
  - Eunpyeong ST. Mary's Hospital, Seoul
  - Severance Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Bundang Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No